CLINICAL TRIAL: NCT01924611
Title: Two Years Survival Rate of Class II ART Restorations in Primary Molars Using Either Rubber Dam or Cotton Rolls.
Brief Title: Two Years Survival Rate of Class II ART Restorations in Primary Molars Using Two Ways to Avoid Saliva Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Thiago Saads Carvalho, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 134/04
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Dental Caries
Keywords: Dental caries; Atraumatic Restorative Technique
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Atraumatic Restorative Technique using cotton rolls.
  Interventions: Procedure: Atraumatic Restorative Technique using cotton rolls
- Experimental Group (Experimental): Atraumatic Restorative Technique using rubber dam.
  Interventions: Procedure: Atraumatic Restorative Technique

INTERVENTIONS:
Procedure: Atraumatic Restorative Technique using cotton rolls — Atraumatic Restorative Technique using cotton rolls.
  Other Names: Atraumatic Restorative Technique
  Arms: Control Group
Procedure: Atraumatic Restorative Technique — Atraumatic Restorative Technique is typically used in Minimally invasive Dentistry.
  This restoration technique is made using only hand instruments and is possible to be carried out in children in schools.
  This particular time, the isolation of the surgical/tooth area was made using rubber dam as saliva barrier.
  Arms: Experimental Group

SUMMARY:
AIM: To evaluate influence of two methods to avoid saliva contamination on the survival rate of atraumatic restorations in primary molars. 232 children, aged between 6-7 years, of both genders, were selected having one primary molar with a proximal dentine lesion. The children were randomly divided into two groups: a control group with class II ART restoration made using cotton rolls and an experimental group using rubber dam. The restorations were made and they were followed up every six months. After two years, the results were compilated and analyzed.

DETAILED DESCRIPTION:
To evaluate influence of two methods to avoid saliva contamination on the survival rate of atraumatic restorations in primary molars. 232 children, aged between 6-7 years, of both genders, were selected having one primary molar with a proximal dentine lesion. The children were randomly divided into two groups: a control group with class II ART restoration made using cotton rolls and an experimental group using rubber dam. The restorations were made and they were followed up every six months. After two years, the results were compilated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders enrolled in school,
* Children aged between 6 and 7 years,
* having cavity with access to ART hand instruments,
* cavity with a mesio-distal maximum dimension of 1mm and a buccal-lingual maximum dimension of 2mm length, measured on the oclusal surface,
* proximal surface of the adjacent tooth should be unimpaired, without visible lesions,

Exclusion Criteria:

* Cavity lesions having pulpal involvement, swelling, fistula or pain were not included in the study,
* Children out of the age range,

Ages: 6 Years to 7 Years | Sex: All
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2004-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of teeth with fractured restorations. | 2 years
  The teeth were assessed every 6 months for a period of 2 years and they were graded according to restoration fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Evert van Amerongen, DDS, PhD, Professor, Study Director — Academic Centre for Dentistry in Amsterdam; Fabio Correia Sampaio, DDS PhD PostDoc, Study Director — UFPB
Locations (1):
- Universidade Federal da Paraíba, João Pessoa, Paraíba, Brazil